CLINICAL TRIAL: NCT02022202
Title: Breast Cancer Genome Guided Therapy Study (BEAUTY)
Acronym: BEAUTY
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC1137; 11-007860 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2024-10-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Invasive Breast Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast cancer tissue and blood specimens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research study is to better understand the reasons why or why not breast cancers are destroyed by standard chemotherapy. This information will be used to develop new and better cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histological confirmation of invasive breast cancer.
* Confirmation of breast cancer lesion ≥ 1.5 cm in size by any clinical (physical examination measurement) or radiographic criteria (mammogram, ultrasound or MRI) in the ipsilateral breast.

  * Note: Benign breast disease, LCIS or DCIS in the contralateral breast is allowed. Contralateral invasive breast cancer is allowed if disease is of clinically lower stage and the higher stage lesion will be the study lesion for all biopsies and tissue samples.
  * Note: Disease in axilla only is not eligible.
  * Note: Patients that have a contraindication or inability to have an MRI may still be enrolled on study and not participate in the MRI at any of the study specific time points.
  * Note: For patients with bilateral disease the higher clinical stage disease will be the study lesion that will undergo study biopsies and tissue samples from surgery and the contralateral lesion will NOT undergo research biopsies and tissue samples.
* Men or women who are to begin neoadjuvant chemotherapy for treatment of Stage I-III Her 2 negative breast cancer with paclitaxel followed by either the combination of 5-fluorouracil, epirubicin and cyclophosphamide (FEC) or the combination of doxorubicin and cyclophosphamide (AC). OR Men or women who are to begin neoadjuvant chemotherapy for treatment of Stage I-III Her 2 positive breast cancer with paclitaxel followed by either the combination of 5-fluorouracil, epirubicin and cyclophosphamide (FEC) or the combination of doxorubicin and cyclophosphamide (AC). MC1137 Trastuzumab will be given concurrently with the taxane portion and can be given concurrently with FEC (but not AC) at the discretion of the medical oncologist.

  * Note: Her2 positive disease is defined to be: HER2 score of 3+ by IHC or HER2 gene amplification by FISH.
* Provide informed written consent.
* Willing to return to Mayo Clinic in Rochester, MN, Mayo Clinic in Arizona, or Mayo Clinic in Florida for imaging correlative, surgery, and follow-up.
* Willing to provide blood samples for correlative research purposes.
* Willing to provide tissue samples for correlative research purposes.
* ECOG Performance Status ≤ 2.

Exclusion Criteria:

* Receiving any investigational agent which would be considered as a treatment for the primary neoplasm.
* Other active malignancy ≤ 5 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix.

  * Note: If there is a history or prior malignancy, they must not be receiving any other treatment for their cancer.
* Patients who are not planning to receive neoadjuvant chemotherapy.
* Biopsy proven Stage IV disease.
* Patients who are pregnant or nursing.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2012-03-03 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Goetz, M.D., Study Chair — Mayo Clinic; Donald W. Northfelt, M.D., Principal Investigator — Mayo Clinic campus in Arizona; Judy C. Boughey, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic campus in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Derived] Leon-Ferre RA, Whitaker KR, Suman VJ, Hoskin T, Giridhar KV, Moore RM, Al-Jarrad A, McLaughlin SA, Northfelt DW, Hunt KN, Conners AL, Moyer A, Carter JM, Kalari K, Weinshilboum R, Wang L, Ingle JN, Knutson KL, Ansell SM, Boughey JC, Goetz MP, Villasboas JC. Pre-treatment peripheral blood immunophenotyping and response to neoadjuvant chemotherapy in operable breast cancer. Breast Cancer Res. 2024 Jun 10;26(1):97. doi: 10.1186/s13058-024-01848-z. PMID 38858721
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy
Started | 132 (8 patients withdrew consent prior to beginning neoadjuvant chemotherapy)
Completed | 124
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Disease Progression | 3
Not completed — Desire go to immediately to surgery | 3

BASELINE CHARACTERISTICS:
Arm/Group | Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy
Number analyzed (Participants) | 132
Age, Customized [Count of Participants; unit: Participants]
  Age: <30 | 2
  Age: 30-39 | 21
  Age: 40-49 | 36
  Age: 50-59 | 40
  Age: 60-69 | 24
  Age: 70+ | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 129
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 132
Clinical T-stage [Count of Participants; unit: Participants] — T1 (includes T1a, T1b, and T1c): Tumor is 2 cm (3/4 of an inch) or less across.
  T2: Tumor is more than 2 cm but not more than 5 cm (2 inches) across.
  T3: Tumor is more than 5 cm across.
  T4 (includes T4a, T4b, T4c, and T4d): Tumor of any size growing into the chest wall or skin. This includes inflammatory breast cancer.
  Participants
    T1 | 12
    T2 | 55
    T3 | 60
    T4 | 5
Clinical N-stage [Count of Participants; unit: Participants] — N0: Cancer has not spread to nearby lymph nodes. N1: Cancer has spread to 1-3 axillary (underarm) lymph node(s), and/or cancer is found in internal mammary lymph nodes on sentinel lymph node biopsy.
  N2: Cancer has spread to 4-9 lymph nodes under the arm, or cancer has enlarged the internal mammary lymph nodes.
  N3: Cancer is found in at least one axillary lymph node (with at least one area of cancer spread greater than 2 mm) and has enlarged the internal mammary lymph nodes or cancer has spread to the lymph nodes under the collarbone or above the collarbone on the same side of the cancer
  Participants
    N0 | 56
    N1 | 69
    N2 | 4
    N3 | 3

OUTCOME MEASURES:

1. Primary Outcome: DNA From the Germline and Breast Tumor for the Identification of Novel Somatic Changes Within Gene and Gene Pathways.
Description: To obtain DNA from the germline and breast tumor for the identification of novel somatic changes within gene and gene pathways that are potentially "druggable" in men or women with breast cancer undergoing a standard neoadjuvant paclitaxel (with or without trastuzumab), followed by a standard anthracycline containing regimen (e.g. doxorubicin and cyclophosphamide) for breast cancer. We will report the median frequency and range of mutations observed for 30 mutated genes of interest.
Time Frame: 1 year 3 months
Population: Pre-NAC tumor and germline sequencing data were generated for 122 patients
Measure: Median (Full Range); unit: mutations
Groups:
- Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy (NAC): Patients received12 weeks of weekly paclitaxel (with trastuzumab for human epidermal growth factor receptor 2-positive [HER2+] malignancies), followed by four cycles of an anthracycline-based regimen. Surgery was performed following completion of NAC, and residual cancer burden (RCB) scores were calculated.
Arm/Group | Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy (NAC)
Number analyzed (Participants) | 122
mutations | 3 [1 to 30]

2. Primary Outcome: Frequency of Known Tumor Mutations for Which Current Drug Therapies Already Exist.
Description: To determine the number of patients with one or more known tumor mutations for which current drug therapies already exist (e.g. BRAF, C-KIT, EGFR mutation, KRAS, PTEN, PI3K).
Time Frame: 1 year 3 months
Population: Pre-NAC tumor and germline sequencing data were generated for 122 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy (NAC)
Number analyzed (Participants) | 122
Participants | 78

3. Primary Outcome: Association Between Breast Cancer Events and Patient-derived Xenografts (PDX) Engraftment
Description: Using breast cancer tissue obtained prior to chemotherapy in all patients and following the completion of chemotherapy (in patients with residual tumors > 2 cm or residual nodal disease), to develop tumor xenograft cell lines for mechanistic and functional studies to determine whether mutations identified are associated with the malignant phenotype and response to associated drugs which target the gene and/or pathways. The breast cancer relapse rate of patients that received pre-NAC PDX engraftment will be reported.
Time Frame: 1 year 3 months
Population: 113 patients had pre-NAC PDX engraftment
Measure: Number; unit: percentage of patients
Arm/Group | Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy (NAC)
Number analyzed (Participants) | 113
percentage of patients | 13.6

4. Primary Outcome: Somatic Alterations Identified Are Associated With Pathologic Complete Response to Therapy.
Description: To determine whether somatic alterations identified above are associated with pathologic complete response (pCR) to therapy. The number of patients experiencing a pCR with one or more somatic alterations will be reported.
Time Frame: 1 year 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy (NAC)
Number analyzed (Participants) | 132
Participants | 44

5. Secondary Outcome: 99mTc-sestamibi Uptake and Pathologic Response Following Neoadjuvant Chemotherapy.
Description: Assess the association between changes in 99mTc-sestamibi uptake and pathologic response following neoadjuvant chemotherapy (MCR participants only). Sensitivity, specificity, positive predictive value, and negative predictive value after NAC at MRI and MBI will be reported.
Time Frame: 1 year 3 months
Population: Only patients underwent both MRI and MBI after NAC
Measure: Number; unit: percent
Arm/Group | Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy (NAC)
Number analyzed (Participants) | 90
percent
  Sensitivity for MRI | 69.4
  Positive predictive value for MRI | 81.4
  Negative predictive value for MRI | 71.4
  Sensitivity for MBI | 58.9
  Positive predictive value for MBI | 84.6
  Negative predictive- value for MBI | 54.9

ADVERSE EVENTS:
Description: Adverse events were not collected for this specimen collection trial.
Arm/Group | Individuals Aged 18 or Older With Stage I-III BC Who Plan to Undergo Neo-adjuvant Chemotherapy (NAC)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT02022202/Prot_SAP_000.pdf
  • Informed Consent Form (2014-01-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT02022202/ICF_001.pdf